CLINICAL TRIAL: NCT04170686
Title: Acceptability and Efficacy of the Zemedy App for Irritable Bowel Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: Bold Health Inc. (Industry)
Responsible Party: Principal Investigator, Melissa Hunt, PhD, Associate Director of Clinical Training, University of Pennsylvania
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 833848
Record Dates: First submitted 2019-11-14; First posted 2019-11-20 (Actual); Results first posted 2020-12-24 (Actual); Last update posted 2021-02-16 (Actual); Status verified 2021-01

CONDITIONS: Irritable Bowel Syndrome
Keywords: cognitive behavioral therapy; self-help; irritable bowel syndrome
MeSH Terms: conditions — Irritable Bowel Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate Treatment (Experimental): Participants will have immediate access to the self-help app. They will take 8 weeks to work through the content at their own pace.
  Interventions: Behavioral: Zemedy App for Irritable Bowel Syndrome
- Waitlist Control (No Intervention): Participants in the waitlist will receive no intervention for 8 weeks, other than a few "check in" emails from study personnel. At the end of 8 weeks, they will be crossed over to the active treatment group and will be given access to the app.

INTERVENTIONS:
Behavioral: Zemedy App for Irritable Bowel Syndrome — The Zemedy App for irritable bowel syndrome is designed to be an engaging, self-help app for people with irritable bowel syndrome. It is based on empirically supported cognitive-behavioral, and GI focused hypnotherapy interventions for IBS.
  Arms: Immediate Treatment

SUMMARY:
The purpose of this research is to assess if a new self-help app for IBS is an acceptable and effective intervention for improving the overall quality of life in patients with Irritable Bowel Syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of IBS. Own a smart phone. Speak English

Exclusion Criteria:

* Under age of consent (18) Diagnosed with another GI disorder (e.g. celiac disease, inflammatory bowel disease)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 146 (Actual)
Dates: Start 2019-10-28 (Actual); Primary Completion 2020-09-28 (Actual); Study Completion 2020-09-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Melissa G Hunt, PhD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hunt M, Miguez S, Dukas B, Onwude O, White S. Efficacy of Zemedy, a Mobile Digital Therapeutic for the Self-management of Irritable Bowel Syndrome: Crossover Randomized Controlled Trial. JMIR Mhealth Uhealth. 2021 May 20;9(5):e26152. doi: 10.2196/26152. PMID 33872182

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 146 potential participants were consented and screened. 25 individuals met exclusion criteria (severe depression) and were not randomized.
Groups:
- Immediate Treatment: Participants will have immediate access to the self-help app. They will take 8 weeks to work through the content at their own pace.
  Zemedy App for IBS: The Zemedy App for IBS is designed to be an engaging, self-help app for people with irritable bowel syndrome. It is based on empirically supported cognitive-behavioral, and GI focused hypnotherapy interventions for IBS.
Period: Screening
Arm/Group | Immediate Treatment | Waitlist Control
Started | 74 | 72
Completed | 62 | 59
Not Completed | 12 | 13
Not completed — Physician Decision | 12 | 13
Period: Randomization and Treatment
Arm/Group | Immediate Treatment | Waitlist Control
Started | 62 | 59
Completed | 36 | 44
Not Completed | 26 | 15
Not completed — Lost to Follow-up | 26 | 15

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Immediate Treatment | Waitlist Control | Total
Number analyzed (Participants) | 62 | 59 | 121
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.21 (10.1) | 30.71 (10.2) | 32 (10.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 49 | 42 | 91
  Male | 13 | 17 | 30
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 4 | 1 | 5
  Black or African American | 4 | 2 | 6
  White | 42 | 50 | 92
  Multiple Race or Other | 8 | 3 | 11
  Hispanic | 4 | 3 | 7
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 62 | 59 | 121
Irritable Bowel Syndrome Quality of Life [Mean (Standard Deviation); unit: units on a scale] — Scale scores range from 0-100 with higher scores reflecting more impairment (worse outcome)
  units on a scale | 53.63 (18.67) | 60.48 (18.29) | 56.97 (18.7)
Gastrointestinal Symptom Rating Scale [Mean (Standard Deviation); unit: units on a scale] — Scale scores range from 0-78 with high scores representing worse GI symptoms.
  units on a scale | 36.76 (12.77) | 37.75 (12.02) | 37.42 (12.4)
GI Cognitions Questionnaire [Mean (Standard Deviation); unit: units on a scale] — Scale measures distorted, catastrophic beliefs about the social and occupational implications of having gastrointestinal symptoms. Scale scores range from 0 to 64 with higher scores representing worse outcomes (more distorted, catastrophic beliefs about GI symptoms)
  units on a scale | 36.76 (12.77) | 37.75 (12.02) | 37.24 (12.4)
Visceral Sensitivity Index [Mean (Standard Deviation); unit: units on a scale] — Scale measures anxiety about visceral (gut) sensations. Scale scores range from 0 to 75 with higher scores representing more anxiety.
  units on a scale | 51.74 (12.29) | 53.54 (11.44) | 52.62 (11.9)
Fear of Food Questionnaire [Mean (Standard Deviation); unit: units on a scale] — Scale measures fear of food and eating. Scale scores range from 0-90 with higher scores representing more fear and impairment.
  units on a scale | 52.87 (19.9) | 55.46 (18.2) | 54.13 (19.1)
Patient Health Questionnaire 9 [Mean (Standard Deviation); unit: units on a scale] — The PHQ measures the frequency of the 9 cardinal symptoms of depression. Scale score range from 0-27 with higher scores representing more severe/frequent depressive symptoms.
  units on a scale | 8.32 (5.29) | 11.03 (4.66) | 9.64 (5.16)
Depression Anxiety and Stress Scale - Depression Subscale [Mean (Standard Deviation); unit: units on a scale] — The depression subscale of the Depression Anxiety and Stress Scale (DASS) ranges from 0-42 with higher scores representing worse depression.
  units on a scale | 11.65 (9.88) | 15.59 (10.69) | 13.57 (10.43)
Depression Anxiety and Stress Scale - Stress Subscale [Mean (Standard Deviation); unit: units on a scale] — The Stress subscale of DASS measures emotional reactivity to perceived stress. It ranges from 0-42 with higher scores reflecting more distress.
  units on a scale | 17.84 (9.56) | 18.71 (8.97) | 18.26 (9.25)
Depression Anxiety and Stress Scale - Anxiety Subscale [Mean (Standard Deviation); unit: units on a scale] — The Anxiety subscale of the DASS measures the affective and physical symptoms of anxiety. It ranges from 0-42 with higher scores representing worse anxiety.
  units on a scale | 12.03 (7.35) | 13.19 (9.14) | 12.6 (8.25)

OUTCOME MEASURES:

1. Primary Outcome: Irritable Bowel Syndrome Quality of Life
Description: A self-report measure of health related quality of life (HRQL) in people with irritable bowel syndrome. Scores range from 0 to 100. Higher scores are a worse outcome.
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Immediate Treatment | Waitlist Control
Number analyzed (Participants) | 36 | 44
score on a scale | 34.25 (19.78) | 58.19 (18.53)

2. Primary Outcome: Gastrointestinal Symptom Rating Scale
Description: a self-report measure of GI symptom severity. Scores range from 0 to 78. Higher scores are a worse outcome.
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Immediate Treatment | Waitlist Control
Number analyzed (Participants) | 36 | 44
score on a scale | 27.56 (10.12) | 38.18 (10.79)

3. Secondary Outcome: Visceral Sensitivity Index
Description: self-report measure of anxiety specific to visceral sensations. Scores range from 0 to 75. Higher scores are a worse outcome.
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Immediate Treatment | Waitlist Control
Number analyzed (Participants) | 36 | 44
score on a scale | 38.14 (16.21) | 53.57 (12.37)

4. Secondary Outcome: GI Cognitions Questionnaire
Description: self-report measure of catastrophizing specific to GI symptoms. Scores range from 0 to 64. Higher scores are a worse outcome.
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Immediate Treatment | Waitlist Control
Number analyzed (Participants) | 36 | 44
score on a scale | 22.44 (13.72) | 40.84 (11.23)

5. Secondary Outcome: Fear of Food Questionnaire
Description: self-report measure of fear of food. Scores range from 0 to 90. Higher scores are a worse outcome.
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Immediate Treatment | Waitlist Control
Number analyzed (Participants) | 36 | 44
score on a scale | 41.22 (22.23) | 53.75 (18.08)

6. Secondary Outcome: Patient Health Questionnaire
Description: self-report measure of depressive symptoms. Scores range from 0 to 27. Higher scores are a worse outcome.
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Immediate Treatment | Waitlist Control
Number analyzed (Participants) | 36 | 44
score on a scale | 5.78 (4.2) | 10.32 (4.29)

7. Secondary Outcome: Depression Anxiety and Stress Scale - Depression Subscale
Description: Self-report measure of depressive symptoms. Scores ranges from 0 to 42. Higher scores represent worse outcome.
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Immediate Treatment | Waitlist Control
Number analyzed (Participants) | 36 | 44
score on a scale | 7.83 (7.88) | 15.45 (10.39)

8. Secondary Outcome: Depression Anxiety and Stress Scale - Stress Subscale
Description: The stress subscale measures emotional reactivity to perceived stress. Scores range from 0-42 with higher scores representing worse stress reactivity.
Time Frame: 8 weeks
Population: Treatment completers and waitlist control participants at post-treatment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Immediate Treatment | Waitlist Control
Number analyzed (Participants) | 36 | 44
units on a scale | 12.72 (8.65) | 18.82 (9.99)

9. Secondary Outcome: Depression Anxiety and Stress Scale - Anxiety Subscale
Description: Measures affective and physical symptoms of anxiety. Scores range from 0-42 with higher scores representing worse anxiety.
Time Frame: 8 weeks
Population: Treatment completers and waitlist control participants at post-treatment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Immediate Treatment | Waitlist Control
Number analyzed (Participants) | 36 | 44
units on a scale | 8.67 (6.38) | 12.05 (9.72)

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Immediate Treatment | Waitlist Control
All-Cause Mortality (participants affected / at risk) | 0/62 | 0/59
Serious Adverse Events (participants affected / at risk) | 0/62 | 0/59
Other Adverse Events (participants affected / at risk) | 0/62 | 0/59

LIMITATIONS AND CAVEATS:
As is the case with most internet trials we experienced significant attrition from both arms. In the final publication, multiple imputation will be used to account for missing data and both treatment completer and intent-to-treat results will be reported.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2019-11-15): https://cdn.clinicaltrials.gov/large-docs/86/NCT04170686/Prot_001.pdf